CLINICAL TRIAL: NCT06197386
Title: Reliability and Validity of the Athlete Fear Avoidance Questionnaire in Turkish
Status: Recruiting | Type: Observational
Sponsor: Atılım University (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, NAİME ULUG, Director, Atılım University
Other Study IDs: E-59394181
Record Dates: First submitted 2023-12-23; First posted 2024-01-09 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Athletic Injuries
Keywords: Athlete Fear Avoidance Questionnaire (AFAQ)
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High levels of fear avoidance can lead to chronic pain and disability and can predict rehabilitation time in the sports-related injury population. Therefore, taking fear avoidance into account may be useful in creating the most appropriate and effective rehabilitation plan, thus shortening the time to return to play. The aim of our study is to verify the validity and reliability of the Athlete Fear Avoidance Questionnaire (AFAQ) in Turkish.

DETAILED DESCRIPTION:
Sports injuries are a frequent occurrence that many athletes experience annually. Although sports injuries cause physical pain and disorders, they also have a psychological impact. One common psychological response to sports injuries is the fear of re-injury. Other potential psychological reactions of an injured athlete include anxiety, depression, frustration, tension, and decreased self-esteem. Psychological responses to sports injuries are typically highest immediately after the injury and decrease during the rehabilitation process. However, they often relapse just before returning to sports. If left unaddressed, these heightened psychological responses can impede rehabilitation progress and delay the return to sport.

Currently, there are several scales available to measure an athlete's readiness to return to play, such as the Sports Inventory for Pain and the Injury-Psychological Readiness to Return to Sport Scale. However, it is important to note that some of these surveys were conducted with student populations rather than athletes. Additionally, these scales are designed to be applied at the end of the rehabilitation process. The Athlete Fear Avoidance Questionnaire (AFAQ) was specifically developed to assess fear avoidance or pain-related fear in athletes.

The fear avoidance model was developed to explain how individuals experiencing exaggerated pain perception separate 'pain experience' and 'pain behavior' from the actual pain sensation. High levels of fear avoidance can lead to chronic pain and disability and can predict rehabilitation time in the sports-related injury population. Therefore, considering fear avoidance may be helpful in developing an appropriate and effective rehabilitation plan, ultimately reducing the time required to return to play. The purpose of our study is to validate and assess the reliability of the Athlete Fear Avoidance Questionnaire (AFAQ) in Turkish.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed athlete for at least 5 years, being active in sports and training for the last 1 year, and weekly training intensity of at least 5 hours per week.

Exclusion Criteria:

* It was defined as having a history of visual, mental or systemic disease.

Ages: 15 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: athlete
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | December 23, 2023
  The Pain Catastrophizing Scale (PCS) is a self-report scale used to measure exaggerated negative thoughts and feelings related to pain. It consists of 13 items and each item is scored between 0 (never) and 4 (always). Total score ranges from 0 to 52.
  The PCS consists of 3 subscales:
  Rumination: Anxious and repetitive thoughts about pain. Magnification: Exaggerating the severity and importance of pain. Helplessness: Feelings of helplessness and inability to control pain. PCS shows that there is a relationship between the way we perceive and manage pain and the severity of pain. Higher PCS scores are associated with more pain and greater functional impairment.
Fear-Avoidance Beliefs Questionnaire (FABQ) | December 23, 2023
  It is used to evaluate fear-avoidance behaviors related to work and physical activity, especially in patients with chronic low back pain. It consists of 16 items and 2 subscales. In the 2nd, 3rd, 4th and 5th items of the subscale (FABQfa), which includes fear-avoidance behaviors related to physical activities; The subscale (FABQiş), which includes work-related fear-avoidance behaviors, is questioned in the 6th, 7th, 9th, 10th, 11th, 12th and 15th items. Each item is rated between 0-6 points. Minimum score is 0; The highest score is 24 for FABQ(fa) and 42 for FABQ(business). A high score indicates that the patient has high fear-avoidance behaviors.
Athlete Fear Avoidance Survey | December 23, 2023
  The fear avoidance model was developed to explain the process by which "pain experience" and "pain behavior" are separated from the actual pain sensation in individuals presenting the phenomenon of exaggerated pain perception. High levels of fear avoidance can lead to chronic pain and disability and successfully predict rehabilitation time in the sports-related injury population

CONTACTS AND LOCATIONS:
Overall Officials: Naime Uluğ, PhD., Principal Investigator — ATILIM UNİVERSİTY
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided